CLINICAL TRIAL: NCT07314957
Title: The Role of Lifestyle in Maintaining Health: Biological, Psychological and Social Responses of the Organism to Lifestyle
Brief Title: Impact of Lifestyle on Health Maintenance: A Randomized Controlled Trial
Acronym: LifeHealth-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zadar (Other)
Collaborators: General Hospital Zadar (Other); School of Public Health Andrija Štampar (Unknown); Psychiatric Hospital Ugljan (Individual); Agricultural, Food and Veterinary School Stanko Ožanić (Unknown)
Responsible Party: Principal Investigator, Marija Ljubičić, Assistant Professor, PhD, Department of Health Studies, University of Zadar, Croatia, University of Zadar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IP UNIZD 2025-27040; EU Next Generation NPOO (Other Grant/Funding Number: European Union / Sveučilište u Zadru)
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Syndrome; Inactivity/Low Levels of Exercise; Unhealthy Diet; Unhealthy Alcohol Use; Smoking Behaviors; Stress; Sleep Disorder; Obesity & Overweight; Anxiety; Depressed Mood; Emotional Eating Behaviour
Keywords: Habits; Lifestlye; Nutrition; Phisical activity; Stress; Metabolic syndrome; Mental health; Sleep
MeSH Terms: conditions — Metabolic Syndrome; Smoking; Sleep Wake Disorders; Obesity; Overweight; Anxiety Disorders; Consciousness Disorders; Habits; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This randomized, interventional study evaluates the effects of lifestyle interventions on metabolic, oxidative, and psychological health in adults with overweight or obesity. Participants are randomly assigned to one of two groups: combined lifestyle group (physical activity, nutrition education, stress-resilience training), and control group receiving no interventions. The study uses open-label allocation with parallel groups to assess causality between lifestyle intervention and health outcomes. Randomization is performed using a computerized random generator. Participants' adherence is monitored via smart bracelets tracking heart rate, steps, and sleep. Outcomes, including metabolic parameters, oxidative stress, hormonal responses, anthropometric measures, stress, quality of life, are assessed at baseline and at 3, 6,12, months folow-up.
Who Masked: Participant
Masking Description: No other parties besides participants are masked. Researchers, study staff, and outcome assessors are aware of group assignments due to the nature of the interventions. This open-label design allows proper supervision of physical activity, dietary education, and stress-resilience training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Adults aged 20 years and older with overweight or obesity (BMI ≥25 kg/m²), stable body weight over the past 6 months and be physically inactive.
- Lifestyle intervention group (Experimental): Adults aged 20 years and older with overweight or obesity (BMI ≥25 kg/m²), stable body weight over the past 6 months and be physically inactive..
  Interventions: Behavioral: Intervention of physical activity; Behavioral: Mediterranean Diet Education; Behavioral: Behavioral: Stress-Resilience Training

INTERVENTIONS:
Behavioral: Intervention of physical activity — The intervention combines supervised physical activity (2 times a week for 12 weeks) with the use of a smart bracelet to continuously monitor heart rate, steps and hours of sleep. The intervention aims to reduce sedentary behavior and improve metabolic, oxidative and psychological health in adults with overweight or obesity.
  Arms: Lifestyle intervention group
Behavioral: Mediterranean Diet Education — Participants will take part in a 12 week nutritional intervention, followed by a 12 month follow-up period. The program includes 14 weekly group education sessions and one 30-minute individual consultation. Group sessions cover healthy eating principles, Mediterranean diet, intuitive eating, meal planning, hunger and satiety awareness, emotional triggers, mindful eating, real-life nutrition situations, motivation, and strategies for maintaining healthy habits. The individual consultation addresses personal challenges and tailors dietary guidance to the participant's lifestyle and health status. Dietary intake is monitored using structured 24-hour recalls at multiple time points throughout the intervention and follow-up periods.Participants will wear smart bracelets to monitor physical activity, heart rate, and sleep to track their daily routine and progress.
  Arms: Lifestyle intervention group
Behavioral: Behavioral: Stress-Resilience Training — Participants will take part in a 12-week program focused on strengthening psychological resilience and stress management. The program includes workshops and group support sessions to encourage experience sharing and motivation, with additional online and telephone support. Participants will wear smart bracelets to monitor physical activity, heart rate, and sleep to track their daily routine and progress.
  Arms: Lifestyle intervention group

SUMMARY:
This study aims to evaluate the impact of public health interventions on changes in healthy lifestyle habits over time and their subsequent effects on health outcomes. The investigators hypothesize that exposing at-risk populations to structured physical activity programs, education on healthy nutrition, promotion of the Mediterranean diet, and workshops focused on strengthening psychological resilience will lead to improvements in anthropometric, oxidative, metabolic, and psychological parameters. Anthropometric and laboratory measures will be collected at multiple time points throughout the study. The longitudinal follow-up will span 12 months. It is anticipated that sustained adherence to healthy lifestyle behaviors will result in positive lifestyle changes and enhanced health-related quality of life.

DETAILED DESCRIPTION:
Contemporary lifestyle patterns are characterized by a fast pace of life, exposure to stressful stimuli, and unhealthy habits. Physically inactive adults who are exposed to stress, smoke, and have poor dietary habits are at increased risk of developing metabolic syndrome, oxidative stress, overweight, hormonal imbalance, insulin resistance, impaired mental health, and lower health-related quality of life.

Studies confirm that lifestyle is one of the most influential modifiable factors in disease development. This study aims to evaluate whether a structured lifestyle intervention, including supervised physical exercise, adherence to a healthy diet, and stress-resilience training, can improve metabolic health, reduce oxidative stress, and enhance mental health and quality of life in adults with overweight, compared to a control group receiving standard lifestyle advice. Participants will be randomly assigned to one of two groups: supervised lifestyle group with exercise , Mediterranean diet education , stress-resilience and support; and control group receiving standard lifestyle recommendations. Participants in the experimental groups will engage in regular physical activity, follow a Mediterranean diet, participate in psychological resilience-building workshops and support groups, and attend weekly individual and group sessions, followed by a 12-month follow-up period.

The study will assess anthropometric measures (body weight, waist and hip circumference), metabolic parameters (blood glucose, HbA1c, cholesterol, HOMA-IR), oxidative stress markers (AGEs), hormonal responses (cortisol, thyroid hormones), mental health, perceived stress, and quality of life. Participants will wear smart bracelets to monitor daily activity, steps, heart rate, and sleep. Measurements will be taken at baseline, immediately after the 12-week intervention (3 month), and during follow-up at 6, and 12 months.

The investigators hypothesize that the structured lifestyle intervention combining physical activity, Mediterranean diet education, and stress-resilience training will lead to significant improvements in metabolic, oxidative, and psychological health outcomes compared to standard lifestyle advice.

The scientific findings gained from this study may significantly contribute to understanding the effectiveness of lifestyle interventions in preventing chronic diseases associated with unhealthy lifestyles. The findings from this study are expected to provide insights into effective lifestyle interventions for at-risk populations, ultimately benefiting both individuals and communities. These interventions can improve the effectiveness of programs aimed at preventing the development of metabolic and chronic diseases, thereby enhancing overall health and quality of life. In addition, the results are anticipated to contribute to evidence-based public health policies and inform strategies for the prevention and management of chronic non-communicable diseases.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 20 years and older
* overweight or obesity (BMI ≥25 kg/m²),
* stable body weight over the past 6 months
* physically inactive.

Exclusion Criteria:

* HbA1c >12%
* insulin therapy
* severe psychiatry and severe chronic illnesses of parents
* diseases of the hypothalamus and pituitary and adrenal gland
* mobility restriction
* tetraplegia
* use of obesity pharmacotherapy
* malignant disease and chemotherapy
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mediterranean diet adherence | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Assessed using validated dietary questionnaires to evaluate participants' adherence to Mediterranean diet principles and monitor changes over time.
  The Mediterranean Dietary Serving Score (MDSS) evaluates 14 food groups, including cereals, fruits, vegetables, olive oil, nuts, dairy, meat, fish, eggs, legumes, potatoes, wine/beer, and sweets. Consumption is rated on a 7-point Likert scale. Scores above 14 indicate regular adherence to a Mediterranean diet.
Physical Activity | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Assessed using the Godin Leisure-Time Exercise Questionnaire to evaluate participants' frequency and intensity of physical activity during free time, and to monitor changes in exercise behavior over time.
  Godin Leisure-Time Exercise Questionnaire (GLTEQ), calculates a total score by multiplying the weekly frequency of strenuous, moderate, and light activities by 9, 5, and 3, respectively. Higher scores indicate greater levels of physical activity and allow monitoring of changes in exercise behavior over time.
Sleep Hygiene | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Assessed using validated sleep hygiene questionnaires to evaluate participants' sleep habits, routines, and behaviors that promote restorative sleep.
  The Sleep Hygiene Index (SHI) consists of 13 items for self-assessment of sleep-related behaviors. Participants rate how often they engage in specific behaviors on a 5-point scale: 0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = always. Scores are summed to provide a global sleep hygiene score, with higher scores indicating poorer (maladaptive) sleep hygiene and a greater presence of behaviors that disrupt sleep quality
Perceived Stress | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Self-reported questionnaire to assess perceived stress levels. The Perceived Stress Scale-10 (PSS-10) assesses the perception of stressful situations over the past month through 10 items rated on a 0-4 scale. Total scores range from 0 to 40, with higher scores indicating higher perceived stress levels.
Healthy Days (Physical and Mental Health) | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Assessed using the CDC Healthy Days questionnaire to evaluate the number of days in the past 30 days when participants perceived their physical or mental health as not good.
  The Health Related Quality of Life 14 item measure (CDC HRQOL 14) is a generic self report questionnaire developed by the U.S. Centers for Disease Control and Prevention to assess overall health related quality of life. It comprises 14 items that capture perceived physical and mental health status over the past 30 days, including self rated general health, the number of days with poor physical health, poor mental health, days when health limited usual activities, and additional questions on activity limitations and symptoms such as pain, depression, anxiety, rest, and energy. The measure provides a summary of health related quality of life and has been widely used in public health surveillance, research, and population health studies. Higher scores generally reflect poorer health related quality of life.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Calculated from measured weight and height to assess changes in body composition.
  Body weight will be measured using a Tanita scale. Body Mass Index (BMI) will be calculated by dividing body weight in kilograms by the square of body height in meters (kg/m²). Reference values will be applied: 18.5-24.9 kg/m² as normal weight, 25-29.9 kg/m² as overweight, and ≥30 kg/m² as obesity.
HbA1c | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Measured from capillary blood using a point-of-care device to assess long-term changes in blood glucose control following lifestyle interventions.
  HbA1c will be measured from capillary blood samples and expressed as a percentage (%) or in mmol/mol. Reference values will be applied, with 4-5.6 % (20-38 mmol/mol) considered normal, 5.7-6.4 % (39-46 mmol/mol) indicating prediabetes, and ≥6.5 % (≥48 mmol/mol) indicating diabetes.
Waist Circumference | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Waist circumference will be measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest using a flexible measuring tape. Reference values will be applied: <94 cm for men and <80 cm for women as normal, 94-102 cm for men and 80-88 cm for women as increased risk, and >102 cm for men and >88 cm for women as high risk of metabolic complications.
Advanced Glycation End Products (AGEs) | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Advanced Glycation End Products (AGEs) will be measured non-invasively in the skin using an AGE Reader device as a marker of oxidative stress. Skin autofluorescence will be assessed on the forearm of the participant's dominant arm, placed on the armrest of the AGE Reader device (DiagnOptics, Groningen, Netherlands). After entering the participant's age, the device displays the AGEs result in arbitrary units (AU). Reference values for advanced glycation end products (AGEs) will be age-dependent. For ages 20-30 years, the reference value is 1.53 ± 0.30 AU; for 30-40 years, 1.73 ± 0.42 AU; for 40-50 years, 1.81 ± 0.36 AU; for 50-60 years, 2.09 ± 0.36 AU; for 60-70 years, 2.46 ± 0.57 AU; for 70-80 years, 2.73 ± 0.55 AU; and for participants aged ≥80 years, 2.71 ± 0.44 AU.
Lipid Profile (Total Cholesterol, LDL, HDL, Triglycerides) | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Measured from fasting blood samples to assess cardiovascular risk. Reference values will be applied, with total cholesterol <5.0 mmol/L, LDL <3.0 mmol/L, HDL ≥1.0 mmol/L for men and ≥1.2 mmol/L for women, and triglycerides <1.7 mmol/L considered within the normal range.
HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Calculated from fasting glucose and insulin to evaluate insulin resistance. Reference values will be applied, with HOMA-IR <2.5 considered normal, 2.5-3.9 indicating moderate insulin resistance, and ≥4.0 indicating significant insulin resistance.
Salivary Cortisol | Baseline, 3 months after intervention
  Collected at four time points during the day to evaluate stress response and HPA axis function.
  Salivary cortisol will be measured at four time points during one day: immediately upon awakening, 30 minutes after awakening, at 16:00, and at 22:00. Salivary cortisol will be measured in nmol/L. Reference values are ≤19 nmol/L for morning cortisol and ≤8 nmol/L for evening cortisol.
Psychological Resilience | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Self-reported questionnaire to assess participants' coping capacity. The Brief Resilience Scale (BRS) is a short questionnaire with 6 questions, used for the assessment of an individual's ability to recover from stress, where a higher score denotes higher stress resilience (average score <3.0 equals low, and score >4.3 denotes high resilience)
Mental Health - The Generalized Anxiety Disorder Scale (GAD-7) | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  Assessed using validated self-report questionnaires to evaluate symptoms of depression and anxiety and monitor changes over time.
  The Generalized Anxiety Disorder Scale (GAD-7) was developed to assess nervous, anxious, and irritable feelings as well as problems with relaxing during the last 2 weeks. A score of 0-4 represents none to minimal level of anxiety, 5-9 is mild level, score of 10-14 indicates moderate level, while a score of 15-21 indicates a severe anxiety level.
Mental Health -The Patient Health Questionnaire (PHQ-9) | Baseline, 3 months after intervention, 6 months after intervention, and 12 months after intervention
  The Patient Health Questionnaire (PHQ-9) was used for the assessment of the presence and severity of depression over the last 2 weeks. Scores of 0-4 represent none to minimal depression, 5-9 represent mild, 10-14 is moderate level of depression, while a score of 15-19 denotes moderate severe, and 20-27 indicates severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zadar, Zadar, Croatia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and confidentiality, as well as to comply with ethical approvals and informed consent agreements. Data contain sensitive personal and health information, and sharing could potentially risk participants' anonymity.

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Stalder T, Kirschbaum C, Kudielka BM, Adam EK, Pruessner JC, Wust S, Dockray S, Smyth N, Evans P, Hellhammer DH, Miller R, Wetherell MA, Lupien SJ, Clow A. Assessment of the cortisol awakening response: Expert consensus guidelines. Psychoneuroendocrinology. 2016 Jan;63:414-32. doi: 10.1016/j.psyneuen.2015.10.010. Epub 2015 Oct 20. PMID 26563991
- [Background] Amanat S, Sinaei E, Panji M, MohammadporHodki R, Bagheri-Hosseinabadi Z, Asadimehr H, Fararouei M, Dianatinasab A. A Randomized Controlled Trial on the Effects of 12 Weeks of Aerobic, Resistance, and Combined Exercises Training on the Serum Levels of Nesfatin-1, Irisin-1 and HOMA-IR. Front Physiol. 2020 Oct 16;11:562895. doi: 10.3389/fphys.2020.562895. eCollection 2020. PMID 33178035
- [Background] Jaacks LM, Sher S, Staercke C, Porkert M, Alexander WR, Jones DP, Vaccarino V, Ziegler TR, Quyyumi AA. Pilot randomized controlled trial of a Mediterranean diet or diet supplemented with fish oil, walnuts, and grape juice in overweight or obese US adults. BMC Nutr. 2018;4:26. doi: 10.1186/s40795-018-0234-y. Epub 2018 May 31. PMID 30271610
- [Background] Leemann L, Martelin T, Koskinen S, Härkänen T, Isola AM. Development and Psychometric Evaluation of the Experiences of Social Inclusion Scale. J Hum Dev Capab 2022;23:400-24. https://doi.org/10.1080/19452829.2021.1985440.
- [Background] Canty-Mitchell J, Zimet GD. Psychometric properties of the Multidimensional Scale of Perceived Social Support in urban adolescents. Am J Community Psychol. 2000 Jun;28(3):391-400. doi: 10.1023/A:1005109522457. PMID 10945123
- [Background] Mastin DF, Bryson J, Corwyn R. Assessment of sleep hygiene using the Sleep Hygiene Index. J Behav Med. 2006 Jun;29(3):223-7. doi: 10.1007/s10865-006-9047-6. Epub 2006 Mar 24. PMID 16557353
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Rosenberg M. Society and the adolescent self-image. Princeton, NJ: Princeton University Press.; 1965.
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Monteagudo C, Mariscal-Arcas M, Rivas A, Lorenzo-Tovar ML, Tur JA, Olea-Serrano F. Proposal of a Mediterranean Diet Serving Score. PLoS One. 2015 Jun 2;10(6):e0128594. doi: 10.1371/journal.pone.0128594. eCollection 2015. PMID 26035442
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Ouanes S, Popp J. High Cortisol and the Risk of Dementia and Alzheimer's Disease: A Review of the Literature. Front Aging Neurosci. 2019 Mar 1;11:43. doi: 10.3389/fnagi.2019.00043. eCollection 2019. PMID 30881301
- [Background] You A, Li Y, Shen C, Fan H, He J, Liu Z, Xue Q, Zhang Y, Zheng L. Associations of non-traditional cardiovascular risk factors and body mass index with metabolic syndrome in the Chinese elderly population. Diabetol Metab Syndr. 2023 Jun 16;15(1):129. doi: 10.1186/s13098-023-01047-4. PMID 37322514
- [Background] Ljubičić M, Matek Sarić M, Klarin I, Rumbak I, Colić Barić I, Ranilović J, et al. Motivation for health behaviour: A predictor of adherence to balanced and healthy food across different coastal Mediterranean countries. J Funct Foods 2022;91:105018. https://doi.org/10.1016/J.JFF.2022.105018.
- [Background] Ljubicic M, Matek Saric M, Klarin I, Rumbak I, Colic Baric I, Ranilovic J, Dzelalija B, Saric A, Nakic D, Djekic I, Korzeniowska M, Bartkiene E, Papageorgiou M, Tarcea M, Cernelic-Bizjak M, Klava D, Szucs V, Vittadini E, Bolhuis D, Guine RPF. Emotions and Food Consumption: Emotional Eating Behavior in a European Population. Foods. 2023 Feb 17;12(4):872. doi: 10.3390/foods12040872. PMID 36832947
- [Background] Gomez-Sanchez L, Gomez-Sanchez M, Tamayo-Morales O, Lugones-Sanchez C, Gonzalez-Sanchez S, Marti-Lluch R, Rodriguez-Sanchez E, Garcia-Ortiz L, Gomez-Marcos MA. Relationship between the Mediterranean Diet and Metabolic Syndrome and Each of the Components That Form It in Caucasian Subjects: A Cross-Sectional Trial. Nutrients. 2024 Jun 19;16(12):1948. doi: 10.3390/nu16121948. PMID 38931300
- [Background] Viscogliosi G, Ettorre E, Chiriac IM, Andreozzi P, Cacciafesta M. Mediterranean Dietary Pattern Adherence and Plasma Lipids Profile. J Endocrinol Diabetes Obesity,;2(2)1-4 2014;2:1-4. https://doi.org/10.47739/1022.
- [Background] Caplin A, Chen FS, Beauchamp MR, Puterman E. The effects of exercise intensity on the cortisol response to a subsequent acute psychosocial stressor. Psychoneuroendocrinology. 2021 Sep;131:105336. doi: 10.1016/j.psyneuen.2021.105336. Epub 2021 Jun 18. PMID 34175558
- [Background] Smaga I, Niedzielska E, Gawlik M, Moniczewski A, Krzek J, Przegalinski E, Pera J, Filip M. Oxidative stress as an etiological factor and a potential treatment target of psychiatric disorders. Part 2. Depression, anxiety, schizophrenia and autism. Pharmacol Rep. 2015 Jun;67(3):569-80. doi: 10.1016/j.pharep.2014.12.015. Epub 2015 Jan 5. PMID 25933971
- [Background] Mehdi S, Wani SUD, Krishna KL, Kinattingal N, Roohi TF. A review on linking stress, depression, and insulin resistance via low-grade chronic inflammation. Biochem Biophys Rep. 2023 Nov 1;36:101571. doi: 10.1016/j.bbrep.2023.101571. eCollection 2023 Dec. PMID 37965066
- [Background] Ljubicic M, Bakovic L, Coza M, Pribisalic A, Kolcic I. Awakening cortisol indicators, advanced glycation end products, stress perception, depression and anxiety in parents of children with chronic conditions. Psychoneuroendocrinology. 2020 Jul;117:104709. doi: 10.1016/j.psyneuen.2020.104709. Epub 2020 May 19. PMID 32450487
- [Background] van Waateringe RP, Fokkens BT, Slagter SN, van der Klauw MM, van Vliet-Ostaptchouk JV, Graaff R, Paterson AD, Smit AJ, Lutgers HL, Wolffenbuttel BHR. Skin autofluorescence predicts incident type 2 diabetes, cardiovascular disease and mortality in the general population. Diabetologia. 2019 Feb;62(2):269-280. doi: 10.1007/s00125-018-4769-x. Epub 2018 Nov 21. PMID 30460578
- [Background] Moldogazieva NT, Mokhosoev IM, Mel'nikova TI, Porozov YB, Terentiev AA. Oxidative Stress and Advanced Lipoxidation and Glycation End Products (ALEs and AGEs) in Aging and Age-Related Diseases. Oxid Med Cell Longev. 2019 Aug 14;2019:3085756. doi: 10.1155/2019/3085756. eCollection 2019. PMID 31485289
- [Background] Oster H, Chaves I. Effects of Healthy Lifestyles on Chronic Diseases: Diet, Sleep and Exercise. Nutrients. 2023 Oct 31;15(21):4627. doi: 10.3390/nu15214627. PMID 37960280
- [Background] Gerber M, Imboden C, Beck J, Brand S, Colledge F, Eckert A, Holsboer-Trachsler E, Puhse U, Hatzinger M. Effects of Aerobic Exercise on Cortisol Stress Reactivity in Response to the Trier Social Stress Test in Inpatients with Major Depressive Disorders: A Randomized Controlled Trial. J Clin Med. 2020 May 11;9(5):1419. doi: 10.3390/jcm9051419. PMID 32403243
- [Background] Park DY, Lee O, Lee YH, Lee CG, Kim YS. Relationship between Change in Physical Activity and Risk of Metabolic Syndrome: A Prospective Cohort Study. J Obes Metab Syndr. 2024 Jun 30;33(2):121-132. doi: 10.7570/jomes24007. Epub 2024 Jun 10. PMID 38852947